CLINICAL TRIAL: NCT01035021
Title: Effect of Neuromuscular Blockade on the Insertion of ProSeal™ Laryngeal Mask Airway and Postoperative Pharyngolaryngeal Discomfort
Brief Title: Neuromuscular Block in Laryngeal Mask Airway(LMA) Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Dr., Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LMA_M_relax
Record Dates: First submitted 2009-12-17; First posted 2009-12-18 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: General Anesthesia; Breast Disease
MeSH Terms: conditions — Breast Diseases | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group N (Active Comparator): Anesthesia is induced with propofol and remifentanil and LMA is inserted by the standard technique according to eht manufacturer's instruction. Rocuronium is administered for the operation.
  Interventions: Drug: use of rocuronium when the LMA is inserted
- group R (Active Comparator): Anesthesia is induced with a propofol and remifentanil and rocuronium 0.06 mg/kg is injected. Insertion of LMA is performed by the standard technique according to the manufacturer's instruction.
  Interventions: Drug: use of rocuronium when the LMA is inserted

INTERVENTIONS:
Drug: use of rocuronium when the LMA is inserted — Anesthesia is induced with a propofol and remifentanil in both groups, however rocuronium 0.06 mg/kg is injected only in group R. Insertion of LMA is performed by the standard technique according to the manufacturer's instruction. In group N, rocuronium is administered for the operation.
  Other Names: esmeron

SUMMARY:
The aim of this study is to evaluate the success rate, insertion time and complication depending on the use of neuromuscular blocking agent when inserting the laryngeal mask airway (LMA).

ELIGIBILITY:
Inclusion Criteria:

* 18-70 year
* american society of anesthesiologist status 1-2
* elective general anesthesia

Exclusion Criteria:

* known or predicted difficult airway
* recent sore throat
* mouth opening less than 2.5 cm
* at risk of aspiration

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
success rate and insertion time | when laryngeal mask airway is inserted

SECONDARY OUTCOMES:
complication after the remove of LMA - bleeding, sore throat | 1 hour after the LMA is removed

CONTACTS AND LOCATIONS:
Overall Officials: Hyoseok Na, Pf, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Na HS, Jeon YT, Shin HJ, Oh AY, Park HP, Hwang JW. Effect of Paralysis at the Time of ProSeal Laryngeal Mask Airway Insertion on Pharyngolaryngeal Morbidities. A Randomized Trial. PLoS One. 2015 Aug 7;10(8):e0134130. doi: 10.1371/journal.pone.0134130. eCollection 2015. PMID 26252522